CLINICAL TRIAL: NCT01799265
Title: Transcend Auto vs Commercially Available Device Clinical Evaluation for Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somnetics International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 800383
Record Dates: First submitted 2013-02-19; First posted 2013-02-26 (Estimated); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2022-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; OSA; AutoPAP; PAP; sleep disordered breathing; CPAP; Apnea hypopnea index; AHI
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcend followed by REMstar (Active Comparator): The patient will receive treatment with Transcend during the first night sleep study, followed by treatment with the REMstar on the second night.
  Interventions: Device: Somnetics Transcend Auto; Device: Respironics REMstar Auto with C-Flex
- REMstar followed by Transcend (Active Comparator): The patient will receive treatment with REMstar during the first night sleep study followed by treatment with Transcend on the second night.
  Interventions: Device: Somnetics Transcend Auto; Device: Respironics REMstar Auto with C-Flex

INTERVENTIONS:
Device: Somnetics Transcend Auto
Device: Respironics REMstar Auto with C-Flex

SUMMARY:
The purpose of this study is to determine whether the Transcend Auto is as effective in treating obstructive sleep apnea as another device that is already on the market.

DETAILED DESCRIPTION:
This is a prospective, randomized, crossover trial. Patients will be randomized 1:1 to undergo two full night sleep studies with the Transcend Auto and a commercially available device.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older
* Diagnosis of obstructive sleep apnea
* Presently using CPAP or APAP therapy

Exclusion Criteria:

* Central or mixed apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-02-27; Primary Completion 2013-06-10 (Actual); Study Completion 2013-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Powell, PhD RPSGT, Principal Investigator — Sleep Therapy and Research Center
Locations (3):
- United States (3):
  - Northwind Lung Specialists and Sleep Center, Coon Rapids, Minnesota
  - Whitney Sleep Center, Plymouth, Minnesota
  - Sleep Therapy and Research Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sites screened individuals who were appropriate for study inclusion by chart review followed by telephone interview. Patients were then asked to schedule an office visit. If the screened individual met the selection criteria, and was interested in participation, the subject was asked to provide informed consent for participation. Subjects were considered enrolled in the study at the time of consent.
Groups:
- Transcend Auto Then REMstar Auto: Patients underwent first night sleep study with Transcend followed by second night sleep study with REMstar
- REMStar Then Transcend Auto: Patients underwent first night sleep study with REMStar and second night with Transcend Auto
Period: Overall Study
Arm/Group | Transcend Auto Then REMstar Auto | REMStar Then Transcend Auto
Started | 20 (Each patient underwent one night sleep study with each device) | 21
Completed | 17 | 18
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — inadequate sleep study | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Baseline characteristics were collected for all patients and were not analyzed by treatment arm
Arm/Group | All Patients
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Mean Apnea Hypopnea Index (AHI) During Treatment
Description: Apnea hypopnea index (AHI) will be measured during treatment with each of the devices. AHI = (number of apneas + number of hypopneas) / total sleep time in hours. The minimum score is zero. The higher the score, the more severe the sleep apnea. For example, obstructive sleep apnea is defined as an AHI >/= 15. AHI was measured by the devices and independently by a central laboratory.
Time Frame: first and second night sleep study
Measure: Mean (Standard Deviation); unit: AHI
Groups:
- Transcend: This is the result when treated with Transcend
- REMStar: This is the result when treated with REMStar
Arm/Group | Transcend | REMStar
Number analyzed (Participants) | 35 | 35
AHI | 2.1 (2.0) | 2.0 (2.4)
Statistical Analysis 1: Comparison: Transcend vs REMStar; Hypothesis testing for the primary endpoint was conducted using a one-sided test of non-inferiority with the following null and alternative hypotheses at the 0.05 significance level using the MIXED procedure in SAS, version 9.3: H_0:(ϕ_m ) ̂≥6.9 H_A:(ϕ_m ) ̂<6.9 where (ϕ_m ) ̂ is the estimated AHI difference between Transcend Auto and REMstar Auto from the model described in 3.5.1; Test type: Non-Inferiority — The 95% upper limit of the prediction interval was calculated using the formula (μ ) ̂+t_(k-2)^α √((τ^2 ) ̂+〖(SE) ̂(μ ̂ )〗^2 ),where (μ ) ̂is the estimate average AHI across all studies, (τ^2 ) ̂ is the between-study variation, t_(k-2)^α is the critical value for a t-distribution, k is the number of studies in the meta-analysis, and k-2 are the degrees of freedom for the t distribution. Meta-analyzed statistics to compute the prediction interval were (μ ) ̂=5.0, SE(μ ̂ )=0.9, and (τ^2 ) ̂=8.0; p = .05, t-test, 1 sided; A p-value of .05 was used

2. Secondary Outcome: Unanticipated Adverse Device Effects
Description: Patients will be monitored for unanticipated adverse device effects during each sleep study. Patients will not be followed after the second sleep study.
Time Frame: first and second night sleep study
Measure: Count of Participants; unit: Participants
Groups:
- Transcend; REMStar: Unanticipated Adverse Device Effects
Arm/Group | Transcend | REMStar
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

3. Secondary Outcome: Mean Differences Between Polysomnography (PSG) and Device Measures of Apnea Index (AI) and Hypopnea Index (HI)
Description: Mean hypopnea index will be measure during treatment. HI will be measured during treatment with each of the devices. HI = number of hypopneas / total sleep time in hours. The minimum score is zero. The higher the score, the more severe the sleep apnea. For example, obstructive sleep apnea is defined as an AHI >/= 15. HI was measured by the devices and independently by a central laboratory. Results are reported as the Mean Differences between PSG and Device Hypopnea Index. These differences can be reported as negative values.
Time Frame: first and second night sleep study
Population: Hypopnea index (HI)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Transcend: This is the result when patients were treated with Transcend
- REMStar: This is the result when patients were treated with REMStar
Arm/Group | Transcend | REMStar
Number analyzed (Participants) | 35 | 35
units on a scale | -0.7 (2.3) | 0.2 (1.6)

ADVERSE EVENTS:
Time Frame: Patients were not followed after the second sleep study. Documentation of adverse events stopped after the second night's sleep study.
Description: Low level headache-lightheaded.
Groups:
- Transcend: Transcend Arm
- REMStar: REMStar Arm
Arm/Group | Transcend | REMStar
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 1/20 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcend (N=20) | REMStar (N=21)
headache (General disorders) | 1 (1) | 0 (0) — headache and lightheadedness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less